CLINICAL TRIAL: NCT00822497
Title: The Efficacy of Music Therapy Protocols for Decreasing Pain, Anxiety, and Muscle Tension Levels During Burn Debridement: A Prospective Randomized Crossover Trial
Brief Title: Efficacy of Music Therapy Protocols for Burn Debridement
Acronym: MTS1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: The Cleveland Music School Settlement (Other); Kulas Foundation (Other)
Responsible Party: Xueli Tan, MM, MT-BC, The Cleveland Music School Settlement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 99-00147
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Pain Management
Keywords: music therapy; pain; anxiety; muscle tension
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Music-Based Imagery
  Interventions: Behavioral: Music-Based Imagery (MBI)
- 2 (Experimental): Music Alternate Engagement
  Interventions: Behavioral: Music Alternate Engagement (MAE)
- Control (No Intervention): Debridement under standard care with no music therapy interventions

INTERVENTIONS:
Behavioral: Music-Based Imagery (MBI) — MBI is form of music-assisted relaxation with imagery. This protocol is used at the patients' bedside before and after the debridement process.
  Other Names: Music & Imagery
  Arms: 1
Behavioral: Music Alternate Engagement (MAE) — MAE consisted of a menu of music therapy interventions aimed at engaging the patients in music and diverting them away from the debridement process.
  Other Names: Distraction Technique
  Arms: 2

SUMMARY:
The purpose of this prospective, crossover randomized study is to explore the efficacy of two music therapy protocols on pain, anxiety, and muscle tension levels throughout the debridement process in individuals hospitalized with moderate to severe burns.

DETAILED DESCRIPTION:
The study is a prospective, randomized crossover clinical trial conducted on a 14-bed inpatient comprehensive burn care center. The purpose of this study is to investigate the efficacy of Music-Based Imagery (MBI) and Music Alternate Engagement (MAE) for pain and anxiety management for burn patients throughout the debridement process.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted for at least three days (excluding day of admission)
* Patient is at least seven years old
* Patient is able to communicate, i.e. awake and alert
* Patient is oriented

Exclusion Criteria:

* Patient admitted for/less than three days
* Patient under seven years of age
* Patient not able to communicate, i.e. sedated and/or intubated
* Patient is not oriented, i.e. active psychosis, hallucinations, delusions, late-stage Alzheimer's or dementia diagnoses

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pain, Anxiety, Muscle Tension levels | 7 data points before, during, after debridement

SECONDARY OUTCOMES:
Narcotics & Anxiolytics (dosage) | Throughout debridement process

CONTACTS AND LOCATIONS:
Overall Officials: Xueli Tan, MM, MT-BC, Study Chair — The Cleveland Music School Settlement; Richard B. Fratianne, MD, FACS, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Prensner JD, Yowler CJ, Smith LF, Steele AL, Fratianne RB. Music therapy for assistance with pain and anxiety management in burn treatment. J Burn Care Rehabil. 2001 Jan-Feb;22(1):83-8; discussion 82-3. doi: 10.1097/00004630-200101000-00019. PMID 11227691
- [Background] Fratianne RB, Prensner JD, Huston MJ, Super DM, Yowler CJ, Standley JM. The effect of music-based imagery and musical alternate engagement on the burn debridement process. J Burn Care Rehabil. 2001 Jan-Feb;22(1):47-53. doi: 10.1097/00004630-200101000-00010. PMID 11227684